CLINICAL TRIAL: NCT06375317
Title: A Single-center, Single-arm, Exploratory Clinical Study of Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With PD-L1 Plus Regorafenib in the Treatment of Advanced Hepatocellular Carcinoma After Immunotherapy Failure.
Brief Title: HAIC Combined With PD-L1 Plus Regorafenib in the Treatment of Advanced Hepatocellular Carcinoma After Immunotherapy Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yehua Shen (Other)
Responsible Party: Sponsor-Investigator, Yehua Shen, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-HAIC-001
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC Combined with PD-L1 Plus Regorafenib (Experimental)
  Interventions: Drug: PD-L1 inhibitor: Adebrelimab Injection；Regorafenib Tablets

INTERVENTIONS:
Drug: PD-L1 inhibitor: Adebrelimab Injection；Regorafenib Tablets — PD-L1 injection: 20 mg/kg, administered every 3 weeks (Q3W).
  Regorafenib: 80 mg, orally, once daily (qd), continuously for 14 days per cycle, followed by a 7-day rest period, administered every 3 weeks (Q3W).
  FOLFOX regimen: Oxaliplatin 85 mg/m2, Calcium folinate 400 mg/m2, Fluorouracil 400 mg/m2 as an IV bolus, followed by Fluorouracil 1200 mg/m2 infusion over 23 hours, administered every 3 weeks (Q3W) for a total of 6 cycles.
  The above doses are recommended doses.

SUMMARY:
For patients with advanced liver cancer who have progressed after first-line targeted and immunotherapy , there is currently no standard treatment regimen for second-line therapy. this study aims to explore the efficacy and safety of HAIC combined with PD-L1 and Regorafenib in patients with advanced liver cancer who have failed immunotherapy, not only providing new treatment options for second-line therapy of liver cancer, but also laying the foundation for research on the combination of HAIC and PD-L1 inhibitors plus Regorafenib, which has significant scientific research significance and clinical value.

DETAILED DESCRIPTION:
This is A Single-center, Single-arm, Exploratory Clinical Study of Hepatic Arterial Infusion Chemotherapy (HAIC) Combined with PD-L1 Plus Regorafenib in the Treatment of Advanced Hepatocellular Carcinoma After Immunotherapy Failure.

In clinical practice, second-line liver cancer treatment still mainly relies on single-agent therapy, which may not provide additional clinical benefits for patients. On one hand, a real-world multicenter study published by ESMO in 2023 showed that the combination of ICIs and TKIs may still have potential efficacy in patients who progress after first-line targeted therapy for advanced liver cancer. Secondly, the combination of targeted therapy and local hepatic arterial infusion chemotherapy (HAIC) may provide a new opportunity for patients with advanced liver cancer who progress after targeted therapy. On the other hand, unlike PD-1 inhibitors, PD-L1 inhibitors can block the binding ability of PD-L1 with B7.1 on the surface of T cells, which is advantageous for comprehensive T cell activation. At the same time, PD-L1 monoclonal antibody only blocks the binding of PD-L1 with PD-1, preserving the function of PD-L2 and avoiding side effects such as interstitial lung disease (ILD), thus having better safety. Therefore, this study aims to explore the efficacy and safety of HAIC combined with PD-L1 and Regorafenib in patients with advanced liver cancer who have failed immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced HCC confirmed by imaging or histopathological examination based on biopsy specimens and/or surgical pathology;
* Patients who have failed ≥1 line of PD-1/PD-L1 immune checkpoint inhibitor therapy;
* Imaging diagnosis with at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1);
* Expected survival period ≥3 months;
* ECOG performance status of 0-1;
* Child-Pugh score of grade A (i.e., a score of 5 to 6);
* Adequate organ and bone marrow function;
* Male participants and women of childbearing potential must use contraception from the start of the first dose to 3 months after the last dose;
* Expected good compliance and ability to comply with the study requirements.

Exclusion Criteria:

* Previous history of immunotherapy with any of the following:

  1. Any grade 3 or higher immune-related adverse events (irAEs);
  2. Any unresolved grade 2 irAEs;
  3. Any toxicity resulting in permanent discontinuation of prior anti-PD-1/PD-L1 immunotherapy;
  4. Patients assessed as having progressed within ≤3 months during prior immunotherapy.
* Previous treatment with Regorafenib;
* Known allergy to the study drug or any of its excipients;
* Received any of the following treatments or medications prior to the first study treatment:

  1. Major surgery within 28 days prior to treatment initiation (diagnostic tissue biopsy is allowed).
  2. Use of immunosuppressive medications within 7 days prior to treatment initiation, excluding nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e., not exceeding 10 mg/day of prednisone or its equivalent).
  3. Receipt of immunomodulatory drugs (such as thymosin, interferon, interleukins) within 3 weeks prior to treatment initiation.
  4. Receipt of attenuated live vaccines within 28 days prior to treatment initiation.
  5. Receipt of other systemic anticancer therapy within 28 days prior to treatment initiation.
* Known uncontrollable or symptomatic active central nervous system (CNS) metastases;
* Diagnosis of other active malignancies within 2 years prior to study entry, except for locally treated and cured basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, ductal carcinoma in situ of the breast, and papillary thyroid cancer.
* Presence of any active autoimmune disease or history of autoimmune disease with anticipated recurrence;
* Human immunodeficiency virus (HIV) infection or known AIDS, untreated active hepatitis, HBV-DNA >2000 IU/ml with abnormal liver function; hepatitis C or combined HBV and HCV co-infection;
* Within 6 months prior to study entry, experienced:
* Myocardial infarction, severe/unstable angina, NYHA class 2 or higher heart failure, clinically significant ventricular or supraventricular arrhythmias requiring clinical intervention; poorly controlled hypertension;
* History of gastrointestinal bleeding or tendency to gastrointestinal bleeding within the past 6 months;
* Urine protein ≥++ or 24-hour urine protein >1.0g;
* Inability to swallow study drugs, presence of chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis), and factors affecting drug intake and absorption such as intestinal obstruction.
* Pregnant or lactating women, and women of childbearing potential unwilling to adopt effective contraceptive measures;
* Other patients deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | approximately 1years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 1 years
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable
Progression-Free Survival (PFS) | approximately 2 years
  PFS is defined as time from the start of treatment to progression of disease or death
Overall Survival (OS) | approximately 2 years
  From date of include in this research until the date of death from any cause, whichever came first

IPD SHARING:
Plan to Share IPD: Undecided